CLINICAL TRIAL: NCT00384423
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase IIa Study to Assess the Short-Term Effects of PRX-03140 Alone and in Combination With Donepezil in Subjects With Mild Alzheimer's Disease.
Brief Title: Short Term Effects of PRX-03140 in Patients With Mild Alzheimer's Disease Being Treated With Aricept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epix Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRX-CP-018
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; AD; PRX-03140; Dementia; Epix; Predix; Cognition enhancing
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PRX-03140

SUMMARY:
This is a study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of PRX-03140 administered orally once daily for 14 days in subjects with mild Alzheimer's Disease who are using a stable, well-tolerated 10 mg dose of Aricept (donepezil) but continue to experience worsening AD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* At least 60 years old.
* On a stable 10 mg dose of Aricept for at least 90 days and able to take it in the morning.
* Diagnosis of probable Alzheimer's Disease.
* Mild dementia.
* You or your authorized representative provide voluntary written informed consent.
* Not pregnant, planning a pregnancy, or capable of becoming pregnant.

Exclusion Criteria:

* Any other medical condition which, in the opinion of the Investigator, would jeopardize your safety, impact the validity of the study results, or interfere with your ability to complete the study according to the protocol.
* Intolerance to Aricept.
* Dementia other than Alzheimer's type.
* Parkinson's Disease.
* History of seizure or epilepsy.
* History of stroke.
* Participation in another research study within last 30 days.
* Enrollment in any previous research study testing PRX-03140.
* Use of prescription cognitive enhancing medications (except Aricept) or MAO inhibitors within last 4 weeks.
* Use of tobacco products within last 4 weeks.
* Positive blood screen for Hepatitis B surface antigen or Hepatitis C antibody.
* Positive urine screen for alcohol or drugs of abuse or history of drug or alcohol abuse within last 6 months.
* Major surgery within last 4 weeks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PRX-03140 during 2 weeks of treatment.
Electroencephalogram (EEG) changes through 14 days of treatment.

SECONDARY OUTCOMES:
Changes in cognition after 2 weeks of treatment.
Blood concentrations of PRX-03140 and Aricept during 14 days of treatment.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - California Clinical Trials Medical Group, Inc, Paramount, California
  - Southwest CLinical Research, Rancho Mirage, California
  - Pacific Research Network, Inc, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Torrance Clinical Research, Torrance, California
  - Research Center for Clinical Studies, Darien, Connecticut
  - Miami Jewish Home and Hospital for the Aged, Miami, Florida
  - Berma Research, Plantation, Florida
  - Comprehensive NeuroScience, Inc, St. Petersburg, Florida
  - Meridien Research, St. Petersburg, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - J. Gary Booker, MD, Shreveport, Louisiana
  - Neuroscience Research of the Berkshires, Pittsfield, Massachusetts
  - Neurology Specialists, Dayton, Ohio
  - Saint Johns Office Building, Tulsa, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Alliance for Neuro Research, LLC, Greenville, South Carolina